CLINICAL TRIAL: NCT05501795
Title: The Accuracy of Flap Thickness Versus the Pre-determined Surgical Planning Using WaveLight® FS200
Status: Completed | Type: Observational
Sponsor: Stephen Wexler (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor-Investigator, Stephen Wexler, Medical Director and Surgeon, Bismarck Lasik
Organization: Bismarck Lasik (Other)
Other Study IDs: SW-22-001
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Myopia
Keywords: FS200
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- WaveLight® FS200 femtosecond laser: Flap creation with the WaveLight® FS200 femtosecond laser
  Interventions: Device: WaveLight® FS200 femtosecond laser

INTERVENTIONS:
Device: WaveLight® FS200 femtosecond laser — Flap creation with the WaveLight® FS200 femtosecond laser

SUMMARY:
The objective is to evaluate the resultant thickness of the FS200 created LASIK flap compared to plan at the surgical visit.

DETAILED DESCRIPTION:
This study is a Single site, single-arm, prospective, observational study of the accuracy of the intended flap thickness, after successful bilateral LASIK surgery. Subjects will be assessed pre-operatively, operatively and at 1 day post-operatively. Clinical evaluations will include measurement of visual acuity, manifest refraction, and flap thickness, and flap diameter.

ELIGIBILITY:
Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Appropriate candidate for uncomplicated bilateral LASIK surgery
* Gender: Males and Females.
* Age: 18 or older.
* Refractive error range - SE refractive errors up to 0 to -6D with maximum cylinder up to 3.00D
* Stable refractive error <0.50D change in preceding year
* Contact lens wear discontinued 3 days prior to pre-op exam and the procedure
* Pachymetry above 490μm with residual greater than 270μm
* Candidates who, as determined by the investigator, can safely undergo LASIK with a 120μm flap
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Have good general and ocular health, with no pathology that compromises visual acuity (outside of residual refractive error)

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Patients with usual relative and absolute contraindications for LASIK surgery (severe dry eye, recurrent corneal erosion, uncontrolled Glaucoma, collagen vascular disorders, keratoconus or signs of keratoconus, uncontrolled Diabetes, Herpes)
* Pachymetry below 490μm
* Autoimmune or immunodeficiency diseases
* Patients with signs of inability to understand consent for study and procedure planned
* Patients with history of previous ocular surgery

The principal investigator reserves the right to declare a patient ineligible or non- evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older who are interested in and appropriate candidates for LASIK.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wexler, MD, Principal Investigator — Bismarck Lasik
Locations (1):
- Bismarck Lasik, Bismarck, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WaveLight® FS200 Femtosecond Laser
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | WaveLight® FS200 Femtosecond Laser
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Resultant Thickness of the FS200 Created LASIK Flap Compared to Plan at the Surgical Visit.
Time Frame: 1 day postoperative
Population: 116 Eyes of 58 participants
Measure: Mean (Standard Deviation); unit: um
Units Other Than Participants: Eyes
Arm/Group | WaveLight® FS200 Femtosecond Laser
Number analyzed (Participants) | 58
Number analyzed (Eyes) | 116
um | 0.64 (9)

2. Secondary Outcome: The Resultant Diameter of the FS200 Created LASIK Flap Compared to Plan
Time Frame: 1 day postoperative
Population: 116 Eyes of 58 participants
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | WaveLight® FS200 Femtosecond Laser
Number analyzed (Participants) | 58
Number analyzed (Eyes) | 116
mm | 0.02 (0.05)

3. Secondary Outcome: Pre-operative Pachymetry as Measured by the EX500 Versus the Oculus Pentacam
Description: Thickness measurements compared between 2 devices: the EX500 and the Oculus Pentacam
Time Frame: Day 0 (surgical visit)
Population: 116 Eyes of 58 participants
Measure: Mean (Standard Deviation); unit: um
Units Other Than Participants: Eyes
Groups:
- EX500: Pachymetry as measured by the EX500
- Pentacam: Pachymetry as measured by the Oculus Pentacam
Arm/Group | EX500 | Pentacam
Number analyzed (Participants) | 58 | 58
Number analyzed (Eyes) | 116 | 116
um | 555.2 (30.9) | 553.1 (29.4)
Statistical Analysis 1: Comparison: EX500 vs Pentacam; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.1, Standard Deviation 5.8

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | WaveLight® FS200 Femtosecond Laser
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT05501795/Prot_SAP_000.pdf